CLINICAL TRIAL: NCT06967194
Title: Early Beta-Blocker Administration in Patients With ST Segment Elevation Myocardial Infraction and SCAI B Status
Brief Title: Early Beta Blocker Administration in STEMI Patients With SCAI B Status
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLV-0011-25
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: ST Segment Elevation Myocardial Infarction (STEMI); Cardiogenic Shock Post Myocardial Infarction
Keywords: acute MI; stemi; beta blockers
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Metoprolol

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, double-blind cohort study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Patients treated with Metoprolol 25mg
  Interventions: Drug: Metoprolol (MET)
- Placebo (Placebo Comparator): Patients treated with matching placebo
  Interventions: Drug: Plcacebo

INTERVENTIONS:
Drug: Metoprolol (MET) — Administration of metoprolol 25 mg twice daily
  Other Names: metoprolol 25mg
  Arms: Intervention
Drug: Plcacebo — Administration of matching placebo
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This study is looking at how a medication called beta-blockers (metoprolol) affects patients with a heart attack (STEMI) who are in the cardiac intensive care unit.

When patients are admitted to the unit, they will be randomly placed in one of two groups. One group will get the metoprolol medication, and the other will receive a placebo (a harmless pill that looks like the real medication). All other treatments will be the same for both groups.

During the study, which is 72 hours long, patients will be monitored for blood pressure, heart rate, and lactate levels alterations.

The main goal is to see if the medication helps improve patients condition or prevent it from getting worse. patients safety is a top priority, and if needed, the doctors can stop the study at any time if there are concerns.

DETAILED DESCRIPTION:
A prospective, randomized, double-blind cohort study will be conducted on patients with STEMI who are hospitalized in the cardiac intensive care unit and classified as SCAI B at the time of admission by the attending physician. Patients will be identified upon admission to the unit and randomized into two arms - a control group and an intervention group. Randomization will be performed using sealed envelopes. A block randomization model will be used based on LVEF estimation of >40% or ≤40%.

In the intervention group, patients will receive standard beta-blocker treatment, specifically low-dose metoprolol at 25 mg twice daily. In the control group, patients will receive a placebo. All other standard treatments will be identical between the two study groups, in accordance with the unit's treatment protocol and the clinical status of the patients.

As an integral part of this treatment, patients will be continuously monitored for parameters including blood pressure, heart rhythm, and blood lactate levels.

The treatment duration under this protocol will be 72 hours or until the occurrence of the primary outcome, whichever comes first. The primary outcome is defined as progression of the patient's condition to SCAI C, according to accepted criteria, including an increase in lactate levels, a decrease in urine output, or a change in mental status. Per guidelines, every 24 hours, investigators will re-evaluate each patient. If they meet current criteria for beta-blocker administration (SCAI A status and no contraindications), the study drug will be terminated and active metoprolol will be prescribed.

To ensure patient safety, the treating staff will have the option to request unblinding of the patient's allocation at any time. Additionally, after the enrollment of 100 patients (or after one year, whichever comes first), an interim analysis of the data will be conducted to ensure the study remains within established safety parameters.

An echocardiogram and follow-up visit will be performed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ST-segment elevation myocardial infarction (STEMI) confirmed by ECG, clinical signs, and coronary catheterization.
* Post-catheterization patients classified as SCAI B upon admission to the unit, defined by the presence of tachycardia and/or hypotension without signs of hypoperfusion (i.e., normal lactate levels, normal capillary refill, preserved mental status, and adequate urine output >0.5 mL/kg/hour).
* Age 18 years or older.
* Mentally competent to provide informed consent, understand the study procedures, and comply with medical recommendations.

Exclusion Criteria:

* Pregnancy.
* Inability to provide informed consent.
* Evidence of pulmonary edema.
* Bradycardia (heart rate <60 beats per minute).
* PR interval >240 milliseconds.
* Second- or third-degree atrioventricular (AV) block.
* Active asthma.
* Known hypersensitivity to metoprolol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients progressed from SCAI B to SCAI C | 3 days from enrollment
  number of patients who progressed from SCAI B to SCAI C as measured by - Serum lactate levels > mmol/L urinary output > 0.5 ml/kg/hour slow capillary filling Change in mental status

SECONDARY OUTCOMES:
Rate of in-hospital mortality | during index admission - expected up to 7 days
  The mortality rate of patients during index admission
Need for Mechanical ventilation | During index admission - expected up to 7 days
  The rate of patients that will require mechanical ventilation
Minor adverse events | 3 days from enrollment
  minor events including tachyarrhythmia, bradyarrhythmia, AV blocks
Hospitalizion duration | During index admission - expected up to 7 days
  Time of index hospitalization
Ejection fraction at 30 days | 30 days
  Ejection fraction as measured by echocardiography at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yishay Szekely, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
Privacy of participants

REFERENCES:
- [Background] Pizarro G, Fernandez-Friera L, Fuster V, Fernandez-Jimenez R, Garcia-Ruiz JM, Garcia-Alvarez A, Mateos A, Barreiro MV, Escalera N, Rodriguez MD, de Miguel A, Garcia-Lunar I, Parra-Fuertes JJ, Sanchez-Gonzalez J, Pardillos L, Nieto B, Jimenez A, Abejon R, Bastante T, Martinez de Vega V, Cabrera JA, Lopez-Melgar B, Guzman G, Garcia-Prieto J, Mirelis JG, Zamorano JL, Albarran A, Goicolea J, Escaned J, Pocock S, Iniguez A, Fernandez-Ortiz A, Sanchez-Brunete V, Macaya C, Ibanez B. Long-term benefit of early pre-reperfusion metoprolol administration in patients with acute myocardial infarction: results from the METOCARD-CNIC trial (Effect of Metoprolol in Cardioprotection During an Acute Myocardial Infarction). J Am Coll Cardiol. 2014 Jun 10;63(22):2356-62. doi: 10.1016/j.jacc.2014.03.014. Epub 2014 Mar 30. PMID 24694530
- [Background] Roolvink V, Ibanez B, Ottervanger JP, Pizarro G, van Royen N, Mateos A, Dambrink JE, Escalera N, Lipsic E, Albarran A, Fernandez-Ortiz A, Fernandez-Aviles F, Goicolea J, Botas J, Remkes W, Hernandez-Jaras V, Kedhi E, Zamorano JL, Navarro F, Alfonso F, Garcia-Lledo A, Alonso J, van Leeuwen M, Nijveldt R, Postma S, Kolkman E, Gosselink M, de Smet B, Rasoul S, Piek JJ, Fuster V, van 't Hof AWJ; EARLY-BAMI Investigators. Early Intravenous Beta-Blockers in Patients With ST-Segment Elevation Myocardial Infarction Before Primary Percutaneous Coronary Intervention. J Am Coll Cardiol. 2016 Jun 14;67(23):2705-2715. doi: 10.1016/j.jacc.2016.03.522. Epub 2016 Apr 3. PMID 27050189
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654